CLINICAL TRIAL: NCT06012318
Title: Dynamic Follow-up of Symptoms Based on Patient-reported Outcomes in Immunotherapy for Esophageal Cancer: a Prospective Multicentre Cohort Study (SPRING)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Shantou University Medical College (Other); The General Hospital of Southern Theater Command (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Shantou Central Hospital (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Shenzhen Second People's Hospital (Other); Longgang District People's Hospital of Shenzhen (Other); Shenzhen Third People's Hospital (Other); Shenzhen People's Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Professor of Medicine, Guangdong Provincial People's Hospital
Other Study IDs: SPRING
Record Dates: First submitted 2023-07-26; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Cancer; Patient-reported Outcomes; Immunotherapy
Keywords: Esophageal Cancer; Immunotherapy; Patient-reported Outcomes; Symptom item bank
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monoimmunotherapy group
- Chemoimmunotherapy group

SUMMARY:
Immunotherapy shows satisfactory effectiveness and safety in patients with esophageal cancer. Immunotherapy-based regimens have a better survival benefit compared to previous chemotherapy and radiotherapy. Patient-reported outcomes (PRO) provide a reliable assessment of patients' functional status during treatment. However, the spectrum of symptoms in esophageal cancer patients receiving immunotherapy is uncertain, and there are no studies applying the symptom bank based on PRO to the immunotherapy model for esophageal cancer. In this prospective study, the investigators aimed to preliminarily screen for symptoms associated with immunotherapy for esophageal cancer through a systematic literature review and expert evaluation, and build a symptom item bank for esophageal cancer patients receiving immunotherapy. Adverse symptoms in esophageal cancer patients treated with immunotherapy were collected prospectively. The distribution and severity of the symptoms, as well as the trajectory of symptom change were further analyzed to demonstrate the validity and reliability of the symptom item bank. It would refine the spectrum of symptoms for esophageal cancer patients receiving immunotherapy and provide a foundation for assessing the specific symptom burden in patients with esophageal cancer receiving immunotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed resectable, locally advanced, advanced metastatic esophageal cancer
* Having received or undergoing an immunotherapy-based treatment regimen
* Age 18-75 years
* ECOG PS of 0-2
* Adequate organ function
* Life expectancy > 6 months
* Participants are fully informed about the whole study and are willing to sign the informed consent

Exclusion Criteria:

* Absence of immunotherapy regimen, or recieving radiotherapy.
* Presence of primary tumours elsewhere, such as gastric cancer, lung cancer or cervical cancer
* Severe organ function deterioration and intolerance to immunotherapy
* Pregnant or breast-feeding women
* Previous autoimmune disease
* Any other conditions that may affect patients' safety and compliance
* Psychological, family, social and other factors leading to inability to inform consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study is patients with esophageal cancer who have received or are receiving immunotherapy-based regimens in various stages, including resectable, locally advanced, and advanced stages.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and severity of adverse symptoms | Patients were evaluated from the beginning of immunochemotherapy to three weeks after completion of the last immunochemotherapy treatment. The total time for patient evaluation is less than 6 months.
  Incidence and severity of adverse symptoms in esophageal cancer patients treated with immunotherapy

SECONDARY OUTCOMES:
Trajectory of adverse symptoms | Patients were evaluated from the beginning of immunochemotherapy to three weeks after completion of the last immunochemotherapy treatment. The total time for patient evaluation is less than 6 months.
  Trajectory of adverse symptoms in esophageal cancer patients treated with immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No